Official title: The "RIGHT-SCORE" Study: a Preoperative Risk Score for Postoperative Right Ventricular Dysfunction in Adult Cardiac Surgery.

Date of the document: July 20, 2024

**NCT number:** ID not yet assigned

## Data processing and analysis

Statistical analysis and graphical presentation will be performed using Stata so8ware (StataCorp LLC).

Risk factors for RVD will be identified using univariate and multivariate logistic regression models for the construction of a nomogram. Different points will be assigned to each risk factor according to the adjusted odds ratio (AOR) for each, facilitating the creation of a predictive model for the development of RVD. The consistency of the model will be evaluated as in logistic regression. Internal validation will be performed using bootstrap.

Patients with missing essential data (pre- and postoperative echocardiogram, postoperative medical therapy, preoperative history, and type of surgery) will be excluded from the study. Subgroup analyses will be performed by dividing patients according to the type of cardiac surgery performed (valve surgery, coronary artery bypass gra8ing, thoracic aortic surgery, other) to evaluate the influence of risk factors based on the type of surgery performed and the relative risk of each surgical procedure to develop RVD.